CLINICAL TRIAL: NCT05708534
Title: Evolution of CMV Antiviral T-cell Immunity Over the Next Six Months Initiation of Treatment With Belatacept.
Acronym: VIRABEL
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/0432/OB
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-01

CONDITIONS: Kidney Transplant Infection
MeSH Terms: interventions — Abatacept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Belatacept — Switching from anticalcineurins to belatacept in a cohort of kidney transplant recipients seropositive for CMV

SUMMARY:
Belatacept inhibits T cell activation by blocking the costimulatory signal. In kidney transplantation, it limits the use of anticalcineurins while ensuring a satisfactory level of immunosuppression.

DETAILED DESCRIPTION:
The Rouen strategy consists of offering belatacept to kidney transplant patients with clinical and laboratory intolerance to anticalcineurins with histological toxicity. This strategy improves or stabilizes the graft's glomerular filtration rate (GFR) in patients with poor renal function. However, a high incidence of opportunistic infections (12.1%), mainly due to CMV, has been observed in elderly patients with a GFR less than 25 ml/min. Two-thirds of CMV infections occur within one year of belatacept initiation and can be particularly severe and life-threatening for both patients and the graft. These results led to the implementation of systematic 3-month antiviral prophylaxis with valganciclovir upon the introduction of belatacept.

CMV immune control depends primarily on virus-specific effector/memory T cells. The impact of costimulation blockade on certain persistent viral infections has been studied experimentally. It is significant when the infection is established, but appears variable in the chronic phase depending on the virus type. Viral load appears to be a determining factor in the size of the antiviral T cell repertoire and its functions (lymphocyte exhaustion). In the case of CMV, the consequences of blocking costimulation on the specific effector/memory T cell pool are unknown.

The hypothesis of this project is that, under belatacept, the influence of CMV on the immune system induces quantitative changes in the effector/memory T cell pool (inflation or, conversely, contraction) and/or functional exhaustion, likely leading to a loss of control of viral replication. This study therefore proposes to investigate the evolution of the anti-CMV response in terms of amplitude, specificity, and functionality, after the introduction of belatacept in CMV-positive patients.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant follow-up at Rouen University Hospital
* Clinico-biological intolerance to anticalcineurins defined by GFR < 25 mL/min and/or water and sodium overload justifying the prescription of loop diuretics and/or post-transplant diabetes and/or resistant hypertension (requiring at least 3 treatments antihypertensives including a thiazide diuretic to reach an objective ≤ 140/90 mmHg).
* Having performed a graft biopsy < 3 months old finding lesions of fibrous endarteritis ≥ 2 or arteriolar hyalinosis ≥ 2
* Having undergone collegial validation for the initiation of treatment with belatacept combined with 3-month anti-CMV prophylaxis with oral Valganciclovir.
* Absence of contraindication to belatacept
* Patient who has never received belatacept
* Having a positive CMV serological status

Exclusion Criteria:

* Patient with symptomatic infection
* Pregnant or parturient or breast-feeding woman or lack of proven effective contraception
* Person deprived of liberty by an administrative or judicial decision or person placed under legal safeguard / sub-tutorship or curatorship
* Patient participating in another therapeutic trial or having participated in another trial within 1 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of kidney transplant recipients seropositive for CMV
Sampling Method: Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To study the quantitative changes in anti-CMV T-lymphocyte immunity to the IE-1 antigen within 6 months of a switch from anticalcineurin treatment to belatacept in a cohort of kidney transplant recipients seropositive for CMV | 6 months
  Number of interferon gamma-producing T lymphocytes in response to the IE-1 antigen determined by ELISPOT at M0, M3 and M6.

CONTACTS AND LOCATIONS:
Locations (1):
- University Rouen Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No